CLINICAL TRIAL: NCT02360748
Title: A Plant Based High Protein Diet to Improve Nutritional Outcomes in Dialysis Patients
Brief Title: A Plant Based High Protein Diet to Improve Nutritional Outcomes in Peritoneal Dialysis Patients
Acronym: PBPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: Fresenius Medical Care North America (Industry); DaVita, Inc. (Industry); Food Care, Inc. (Industry)
Responsible Party: Principal Investigator, Naseer Khan, MD, MD, Ochsner Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00011136
Record Dates: First submitted 2015-02-03; First posted 2015-02-11 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: End-Stage Renal Disease; Malnutrition
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single (Experimental): Pilot Study in which patients will be adding food items to improve their nutritional status
  Interventions: Dietary Supplement: Plant based high protein food items

INTERVENTIONS:
Dietary Supplement: Plant based high protein food items — Patients will add high protein plant based food items to their diet

SUMMARY:
The study proposes that addition of high protein plant based diet will improve serum albumin as well serum phosphate for patients with End Stage Renal Disease (ESRD) on Dialysis. Patient will be provided additional food items to help improve their nutritional status.

DETAILED DESCRIPTION:
The purpose of this study is to improve the albumin and nutritional status of patient with ESRD on dialysis. Serum albumin is a marker to show how well the patient's overall nutrition is. When albumin level drops it signifies poor outcome in dialysis patients both in terms of complications as well as mortality. Our goal on dialysis is to improve serum albumin level as close to normal as possible. This study intends to also improve phosphorus level by adding high protein sources which are plant based. In this study we intend to add certain plant based food items which are high in protein content. Studies have shown that these particular food items considerably increase serum albumin level but at the same time they are safe as they do not increase the phosphorous levels in kidney patients. Patients will be provided the additional food items and all their nutritional parameters will be monitored at baseline and during the study period of one month

ELIGIBILITY:
Inclusion Criteria:

* ESRD Patients on dialysis with an albumin of <4.0 with the ability to consent and willingness to enroll in the study

Exclusion Criteria:

* Other exclusions include

  * liver cirrhosis,
  * cardiac cirrhosis,
  * dysphagia due to an old Cerebrovascular accident / muscular dystrophy,
  * Hyperkalemia (>5.5)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Nutritional Parameters, bone and mineral metabolism | one month
  albumin will improve on high protein plant based diet; we will measure patients' baseline nutritional parameters which will include serum album; Calcium and phosphate levels and then follow the same parameters on the dietary intervention

SECONDARY OUTCOMES:
Phosphorous measurements will be followed during the course of the study and on completion | one month
  Hyperphosphatemia will improve on plant based high protein diet
Obesity | one month
  On this intervention we will follow patients' weight as a secondary outcome in obese patients

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - OCHSNER, Baton Rouge, Louisiana
  - Davita, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided
Will upload results

REFERENCES:
- [Background] Kalantar-Zadeh K, Gutekunst L, Mehrotra R, Kovesdy CP, Bross R, Shinaberger CS, Noori N, Hirschberg R, Benner D, Nissenson AR, Kopple JD. Understanding sources of dietary phosphorus in the treatment of patients with chronic kidney disease. Clin J Am Soc Nephrol. 2010 Mar;5(3):519-30. doi: 10.2215/CJN.06080809. Epub 2010 Jan 21. PMID 20093346
- [Background] Noori N, Sims JJ, Kopple JD, Shah A, Colman S, Shinaberger CS, Bross R, Mehrotra R, Kovesdy CP, Kalantar-Zadeh K. Organic and inorganic dietary phosphorus and its management in chronic kidney disease. Iran J Kidney Dis. 2010 Apr;4(2):89-100. PMID 20404416
- [Result] Noori N, Kalantar-Zadeh K, Kovesdy CP, Bross R, Benner D, Kopple JD. Association of dietary phosphorus intake and phosphorus to protein ratio with mortality in hemodialysis patients. Clin J Am Soc Nephrol. 2010 Apr;5(4):683-92. doi: 10.2215/CJN.08601209. Epub 2010 Feb 25. PMID 20185606